CLINICAL TRIAL: NCT05286853
Title: A Phase 3 Randomized Controlled Study of REACT in Participants With Type 2 Diabetes and Chronic Kidney Disease (REGEN-016)
Brief Title: A Study of Renal Autologous Cell Therapy (REACT) in Participants With Type 2 Diabetes and Chronic Kidney Disease
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Why Stopped: Rilparencel is eligible for initial FDA/ RMAT approval pathway upon successful completion Phase3 REGEN006 (PROACT1) trial. Discontinued Phase3 REGEN016 (PROACT2) focused on enrollment outside the US and is not required for initial US registration.
Sponsor: Prokidney (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: REGEN-016
Record Dates: First submitted 2022-02-24; First posted 2022-03-18 (Actual); Last update posted 2024-09-25 (Actual); Status verified 2024-07

CONDITIONS: Type 2 Diabetes Mellitus; Chronic Kidney Diseases
Keywords: REACT; Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Renal Insufficiency, Chronic

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Sham Procedure (Sham Comparator): Participants randomized to the Sham Comparator arm will have 2 sham procedures
  Interventions: Procedure: Sham Comparator
- Experimental (REACT injections) (Experimental): Participants randomized to the experimental arm will receive 2 injections of REACT.
  Interventions: Biological: Renal Autologous Cell Therapy (REACT)

INTERVENTIONS:
Biological: Renal Autologous Cell Therapy (REACT) — Participants receiving institutional standard of care will have a kidney biopsy followed by 2 REACT injections into biopsied and non-biopsied contralateral kidneys 3 months (+30 days) apart and will be followed for 5 years (60 months) since last REACT injection.
  Arms: Experimental (REACT injections)
Procedure: Sham Comparator — Participants receiving institutional standard of care will have 2 sham procedures that simulate real biopsy and injection procedure. No tissue is taken during biopsy and nothing is injected into kidney. The second sham procedure will occur 3 months (+30 days) after the first sham procedure. Participants will be followed for 5 years (60 months) since last sham REACT injection.
  Arms: Sham Procedure

SUMMARY:
The purpose of this study is to assess the safety and efficacy (including durability) of up to 2 REACT injections given 3 months (+30 days) apart and delivered percutaneously into biopsied and non-biopsied contralateral kidneys in participants with T2DM and CKD.

DETAILED DESCRIPTION:
Randomized multi-center, blinded intervention, two cohort , study whereby eligible participants will be randomized 1:1, prior to kidney biopsy, to 1 of 2 cohorts. Cohort 1 participants will undergo sham procedures and be followed for 5 years post last simulated injection.. Cohort 2 participants will receive 2 REACT injections 3 months apart (+30 days) and be followed for 5 years post last injection of the investigational product.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is male or female, 30 to 80 years of age on the date of informed consent.
2. The participant has a clinical diagnosis of T2DM in their health record.
3. The participant has a clinical diagnosis of diabetic nephropathy as the underlying cause of renal disease (diagnosis does not have to be confirmed via renal biopsy) in their health record.
4. The participant has a serum glycosylated hemoglobin (HbA1c) less than 10% at the Screening Visit.
5. The participant has a documented clinical diagnosis of an eGFR greater than or equal to 20 and less than or equal to 44 mL/min/1.73m², not requiring renal dialysis.
6. The participant has an urinary albumin-to-creatinine ratio (UACR) of greater than or equal to 300 and less than or equal to 5,000 mg/g.

Exclusion Criteria:

1. The participant has a history of type 1 diabetes mellitus.
2. The participant has a history of renal transplantation.
3. The participant has a mean systolic blood pressure greater than or equal to 140 mmHg and/or mean diastolic blood pressure greater than or equal to 90 mmHg at screening, across 3 measurements while seated.
4. The participant has hemoglobin level less than 10 g/dL and is not responsive to the standard medical intervention for CKD-related anemia prior to randomization.

Ages: 30 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2024-07-17 (Actual); Primary Completion 2024-09-03 (Actual); Study Completion 2024-09-03 (Actual)

PRIMARY OUTCOMES:
Primary Composite Endpoint | up to 60 Months post last injection of the investigational product or the last simulated injection.
  The time from first injection to the earliest of:
  * At least 40% reduction in eGFR, using the 2009 CKD-EPI serum creatinine equation, sustained for 30 days or
  * eGFR <15 mL/min/1.73m² using the 2009 serum creatinine equation, sustained for 30 days and/or chronic dialysis , and/or renal transplant or
  * Renal or cardiovascular death

SECONDARY OUTCOMES:
First Secondary Endpoint: Time to progression of Chronic Kidney Disease | up to 60 Months post last injection of the investigational product or the last simulated injection
  Time to progression of Chronic Kidney Disease
  * At least 40% reduction in eGFR, using the 2009 CKD-EPI serum creatinine equation, sustained for 30 days or
  * eGFR <15mL/min/1.73m² using the 2009 CKD-EPI serum creatinine equation, sustained for 30 days and/or chronic dialysis, and/or renal transplant or or
  * Renal death
Second Secondary Endpoint: Time to End Stage Renal Disease | up to 60 Months post last injection of the investigational product or the last simulated injection
  Time to End Stage Renal Disease
  * eGFR, <15 mL/min/1.73m² using the 2009 CKD-EPI serum creatinine equation, sustained for 30 days. and/or chronic dialysis, and/or renal transplant or
  * Renal death.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Prokidney
Locations (3):
- Spain (3):
  - IMIM Hospital del Mar Medical Research Institute, Barcelona
  - Hospital Universitario Vall D'Hebron, Barcelona
  - Hospital Universitario 12 de Octubre, Madrid

IPD SHARING:
Plan to Share IPD: No